CLINICAL TRIAL: NCT07260175
Title: adIVO - A Phase II Trial of Ivosidenib Maintenance After SOC Adjuvant Chemotherapy in Curative mIDH1 Cholangiocarcinoma
Brief Title: Phase II Study Evaluating Ivosidenib Maintenance After SOC Adjuvant Chemotherapy in Curative mIDH1 Cholangiocarcinoma
Acronym: adIVO
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Institut für Klinische Krebsforschung IKF GmbH at Krankenhaus Nordwest (Other)
Collaborators: Servier Deutschland GmbH (Industry); Servier Affaires Médicales (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: adIVO; 2024-520219-42-00 (EU CTIS Number); AIO-HEP-0125/ass. (Other: AIO); IKF-081 (Other: Frankfurter Institut für Klinische Krebsforschung IKF GmbH)
Record Dates: First submitted 2025-10-02; First posted 2025-12-03 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Cholangiocarcinoma; IDH Mutation
Keywords: mIDH1 cholangiocarcinoma; ivosidenib maintenance; cholangiocarcinoma; R0-resection
MeSH Terms: conditions — Cholangiocarcinoma | interventions — ivosidenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ivosidenib maintenance (Experimental): Ivosidenib maintenance after SOC adjuvant chemotherapy in curative mIDH1 cholangiocarcinoma
  Interventions: Drug: Ivosidenib

INTERVENTIONS:
Drug: Ivosidenib — Ivosidenib (daily 500 mg) maintenance after SOC adjuvant chemotherapy in curative mIDH1 cholangiocarcinoma
  Other Names: Ivosidenib Pill (daily 500 mg)

SUMMARY:
This study trial is a prospective, multicentre, exploratory, single-arm, open-label phase II study to evaluat ivosidenib maintenance after SOC adjuvant chemotherapy in curative mIDH1 cholangiocarcinoma

DETAILED DESCRIPTION:
The primary objective is to assess the efficacy of ivosidenib maintenance directly after adjuvant SOC chemotherapy in curative mIDH1 iCCA. The corresponding endpoint ist 1-year recurrence-free survival rate (RFS@1year), defined as proportion of patients alive with no disease recurrence 1 year after start of maintenance ivosidenib.

The secondary objective is to evaluate further efficacy as well as to assess safety and impact on the quality of life of ivosidenib maintenance directly after adjuvant SOC chemotherapy in curative mIDH1 iCCA. The corresponding endpoint are:

* RFS, defined as time from start of ivosidenib maintenance to the date of disease recurrence or death to any cause
* Time to recurrence (TTR), defined as time from start of ivosidenib maintenance to the date of disease recurrence
* Time to treatment failure (TTF), defined as time from start of ivosidenib maintenance to the date of premature treatment discontinuation from any cause, including disease recurrence, treatment toxicity or death
* Overall survival (OS), defined as time from enrollment to the date of death from any cause
* Safety
* Quality of life using EORTC QLQ-C30 and EORTC QLQ-BIL21 questionnaires

This is a prospective, multi-center, exploratory, single-arm, open-label phase II study.

Patients with curatively resected intrahepatic cholangiocarcinoma with proven IDH1 mutation, without metastatic spread, in the adjuvant situation (R0-resected), who received 6 months of SOC adjuvant treatment and show at least stable disease under this treatment will be enrolled.

All eligible patients will receive ivosidenib (500 mg qd, 28 days). Patients will be treated within the trial for up to 12 months and the treatment response will be assessed every 8 weeks (Q8W ± 7 days) during trial treatment and every 12 weeks (Q12W ± 14 days) during follow-up until recurrence. Overall, patients will be followed up for 48 months after last patient in or until death, withdrawal of consent, or loss to follow-up (whichever occurs first).

ELIGIBILITY:
Inclusion Criteria:

1. Patient* provides signed informed consent.
2. Patient is ≥ 18 years at the time of given informed consent.
3. Patient has histologically documented curatively resected intrahepatic cholangiocarcinoma, without metastatic spread, in the adjuvant situation (R0-resected)
4. Patient has proven IDH1 mutation (IDH1-variant status evaluated locally by certified test on formalin-fixed paraffin-embedded tumor tissue specimen. If local testing for screening is not possible per local standard, tumor tissue samples will be subject to pre-screening via central IDH1 dPCR)
5. Patient finished adjuvant systemic SOC chemotherapy (with regimens allowed per the protocol) directly prior to trial inclusion.
6. Radiologic imaging available that shows that patient is tumor free at the timepoint of enrollment (not older than 6 weeks from the day of inclusion).
7. Patient has ECOG Performance status ≤ 1
8. Hematological, hepatic and renal function parameters adequate to allow targeted therapy with ivosidenib at investigator´s discretion and IB.
9. Patient has adequate coagulability to allow targeted therapy with ivosidenib at investigator´s discretion and IB. Patients receiving warfarin / Phenprocoumon must be switched to low molecular weight heparin and before starting trial-specific.
10. Patient must be willingly to provide liquid biopsy samples, archival tumor tissue samples (if available), and in the event of disease recurrence, re-biopsy samples (if re-biopsy is considered safe for the patient) for the translational research program.
11. Female patients of childbearing potential or male patients with female partners of childbearing potential must agree to remain abstinent (refrain from heterosexual intercourse) or use contraceptive methods that result in a failure rate of <1% per year during the treatment period and for at least 6 months after the last dose of trial treatment. Male patients with a pregnant partner must agree to remain abstinent or to use a condom for the duration of the pregnancy. Female patients of child-bearing potential must have a negative pregnancy test within the last 7 days prior to the start of trial therapy.
12. Patient is willing and able to comply with the protocol (including contraceptive measures) for the duration of the trial including undergoing treatment and scheduled visits and examinations including follow up.

Exclusion Criteria:

1. Patient has a metastatic or R+ resected biliary tract cancer.
2. Patient received previous therapy with an IDH1 inhibitor.
3. Patient has known presence of tumors other than intrahepatic cholangiocarcinoma or a secondary tumor other than squamous or basal cell carcinomas of the skin or in situ carcinomas of the cervix which have been effectively treated. The sponsor decides to include patients who have received curative treatment and have been disease-free for at least 5 years.
4. Simultaneous, ongoing systemic immunotherapy, chemotherapy, or hormone therapy not described in the trial protocol.
5. Patient receives simultaneous treatment with a different anti-cancer therapy other than that provided for in the trial (excluding palliative radiotherapy only for symptom control).
6. Patient has a stage B cirrhosis according to Child-Pugh criteria (or worse) or cirrhosis (of any grade) with a history of hepatic encephalopathy or clinically significant ascites resulting from cirrhosis. Clinically significant ascites is defined as ascites resulting from cirrhosis requiring diuretics or paracentesis.
7. Patient has known allergic / hypersensitive reactions to at least one of the treatment components.
8. Patient has other serious illnesses or medical ailments within the last 12 months prior to the start of the trial.
9. Patient has a known presence of an active, uncontrollable infection.
10. Patient has QTc > 480ms or other factors that, in the discretion of the investigator increase significantly the risk of QT prolongation or arrhythmic events (e.g. heart failure, hypokalemia, family history of long QT syndrome). NOTE: Medications that prolong the QT interval should be avoided, unless they can be transferred to other medication within ≥ 5 half-lives to dosing or unless the medications can be properly monitored during the study. (If equivalent medication is not available, QTc should be closely monitored).
11. Patient has active disseminated intravascular coagulation.
12. Patient has an active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
13. Patient has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial drug.
14. Patient has any other serious concomitant or medical condition that, in the opinion of the investigator, presents a high risk of complications to the patient or reduces the likelihood of clinical effect. NOTE: strong CYP3A4 inducers or sensitive CYP3A4 substrates with narrow therapeutic window should be avoided, unless they can be transferred to alternative medication within at least 5-half lives prior to dosing.
15. Female patient is pregnant or breast feeding or planning to become pregnant within and 6 months after the end of treatment.
16. Patient who has been incarcerated or involuntarily institutionalized by court order or by the authorities.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-11-18 (Actual); Primary Completion 2030-12 (Estimated); Study Completion 2031-12 (Estimated)

PRIMARY OUTCOMES:
recurrence-free survival rate | 1-year
  1-year recurrence-free survival rate (RFS@1year), defined as proportion of patients alive with no disease recurrence 1 year after start of maintenance ivosidenib

SECONDARY OUTCOMES:
recurrence-free survival | at 66 months
  RFS, defined as time from start of ivosidenib maintenance to the date of disease recurrence or death to any cause
Time to recurrence | after 66 months
  Time to recurrence (TTR), defined as time from start of ivosidenib maintenance to the date of disease recurrence
Time to treatment failure (TTF) | at 66 months
  Time to treatment failure (TTF), defined as time from start of ivosidenib maintenance to the date of premature treatment discontinuation from any cause, including disease recurrence, treatment toxicity or death
Overall survival | at 66 months
  Overall survival (OS), defined as time from enrollment to the date of death from any cause
Safety (adverse events) | at 66 months
  frequency of adverse events
Patient´s Quality of life | at 66 months
  Quality of life using EORTC QLQ-C30
Patient´s Quality of Life | at 66 months
  Quality of life using EORTC QLQ-BIL21

CONTACTS AND LOCATIONS:
Overall Officials: Salah Al-Batran, Prof. Dr., Study Director — Frankfurter Institut für Klinische Krebsforschung IKF GmbH; Thorsten Götze, Prof. Dr., Principal Investigator — Krankenhaus Nordwest GmbH
Locations (4):
- Germany (4):
  - Institute for Clinical Cancer Research Krankenhaus Nordwest, Frankfurt
  - Krankenhaus Nordwest, Frankfurt
  - Uniklinikum Jena, Jena
  - Klinikum rechts der Isar TU München, München

IPD SHARING:
Plan to Share IPD: No
No IPD will be shared